CLINICAL TRIAL: NCT03303820
Title: Analysis of the Impact of the Undernutrition on the Cerebral Infarct in Thrombolized Patients
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: ADIT
Record Dates: First submitted 2017-10-02; First posted 2017-10-06 (Actual); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Thrombosis
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Many clinical trials show that 30 to 50 % of the hospitalized patients are undernourished in various degrees. This prevalence didn't change since 15-20 years The fact is that the present undernutrition in the admission deteriorates during the hospitalization.

Besides, the cerebral vascular accident (AVC) complicates the first days, in at least 50 % of the cases, the disorders of the gulp, which are a risk factor of acquired undernutrition. The nutrition holds an important place in the therapeutic coverage of the AVC. Nevertheless, the link between the undernutrition the entrance and the evolution of the AVC is at the moment only little known. The purpose is to study the impact of the undernutrition in the entrance to the hospital (undernutrition previous to the AVC), on the gravity and the evolution

ELIGIBILITY:
Inclusion Criteria:

* patient admitted in hospital for vascular cerebral accident in 2015
* thrombolytic treatment

Exclusion Criteria:

* no thrombolytic treatment
* transcient ischaemic attack

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patient admitted in hospital for vascular cerebral accident in 2015 with thrombolytic treatment
Sampling Method: Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2016-05-27 (Actual); Primary Completion 2017-05-27 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Rankin score | Day 1; last day of hospitalisation
  measurement of Rankin score at the entrance and at the end of hospitalisation

CONTACTS AND LOCATIONS:
Overall Officials: ZUBER Mathieu, Professor, Study Director — GHPSJ
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France